CLINICAL TRIAL: NCT00899769
Title: Serum Biomarkers for Head and Neck Cancer
Brief Title: Biomarkers in Patients With Head and Neck Cancer and in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000546781; P30CA068485 (NIH); VU-VICC-HN-0530; VU-VICC-IRB-050230
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Immunoenzyme Techniques; Chromatography, Liquid; Mass Spectrometry

INTERVENTIONS:
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood, tissue, and saliva in the laboratory from patients with cancer and from healthy volunteers may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers in patients with head and neck cancer and in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate the differences in serum protein profiles with the differences in the number of peptide matches in patients with squamous cell carcinoma of the head and neck and in healthy volunteers.
* Correlate protein levels with the largest difference in peptide matches in sera in these participants.

OUTLINE: This is a prospective study.

Participants undergo blood, tissue, and saliva collection for biological studies. Samples are analyzed for albumin-bound and non-albumin-bound proteins or IgG via liquid chromatography and tandem mass spectrometry (LC-MS-MS), ELISA, proteomic profiling, and protein expression.

PROJECTED ACCRUAL: A total of 50 patients and 50 healthy volunteers will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Diagnosis of squamous cell carcinoma of the head and neck
  * Healthy volunteer matched by sex, race, birth decade, or smoking status (e.g., current smoker, former smoker, or nonsmoker)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Differences in serum protein profiles and differences in the number of peptide matches
Protein levels and the largest difference in peptide matches in sera

CONTACTS AND LOCATIONS:
Overall Officials: Wendell G. Yarbrough, MD, FACS, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee